CLINICAL TRIAL: NCT03442777
Title: Silicone Adhesive Multilayer Foam Dressings as Adjuvant Prophylactic Therapy for Pressure Ulcer (PU) Prevention: a Multicentric Randomised Open Label Parallel Group Medical Device Trial in Hospitalised Patients at Risk of PU Development
Brief Title: Silicone Adhesive Multilayer Foam Dressings to Prevent Pressure Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KCE-16012
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: patients will be allocated to 1 of the 3 study arms based on a 1:1:1 allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Arm 1 (on top of standard of care) (Experimental): Allevyn® brand silicone adhesive multilayer foam dressings
  * Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Smith & Nephew (Allevyn® brand).
  Interventions: Device: Allevyn® brand silicone adhesive multilayer foam dressings
- Study Arm 2 (on top of standard of care) (Experimental): Mepilex® brand silicone adhesive multilayer foam dressings
  * Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Mölnlycke Health care (Mepilex® brand).
  Interventions: Device: Mepilex® brand silicone adhesive multilayer foam dressings
- Study Arm 3 (standard of care) (No Intervention): * Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * No silicone adhesive multilayer foam dressings will be applied on the skin sites of interest for this trial (sacrum, heel right/left, greater trochanter right/left).

INTERVENTIONS:
Device: Allevyn® brand silicone adhesive multilayer foam dressings — Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Smith&Nephew (Allevyn® brand).
  Arms: Study Arm 1 (on top of standard of care)
Device: Mepilex® brand silicone adhesive multilayer foam dressings — Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Mölnlycke Health care (Mepilex® brand).
  Arms: Study Arm 2 (on top of standard of care)

SUMMARY:
The objective of this study is to determine if silicone adhesive multilayer foam dressings applied to the sacrum, heels and greater trochanter in addition to standard prevention reduce pressure ulcer incidence category II, III, IV, Unstageable and Deep Tissue Injury (DTI) compared to standard pressure ulcer prevention alone, in at risk hospitalised patients. In particular, this trial extends previous trial results obtained in ICU setting. Therefore, only a maximum of 25% of patients will be recruited from ICU settings.

The hypothesis is: 'The use of silicone adhesive multilayer foam dressings as adjuvant prophylactic therapy for pressure ulcer prevention is more effective in reducing pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) incidence rate on sacrum, heels and greater trochanter, compared to standard pressure ulcer prevention alone.' The null hypothesis is: 'The use of silicone adhesive multilayer foam dressings as adjuvant prophylactic therapy for pressure ulcer prevention is not more effective in reducing pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) incidence rate on sacrum, heels and greater trochanter, compared to standard pressure ulcer prevention alone.

DETAILED DESCRIPTION:
A multicentre randomised controlled open label parallel group medical device trial in approximately 8 hospitals in Belgium.

Patients will be randomly allocated to three study arms based on a 1:1:1 allocation:

Study arm 1 (on top of standard of care):

* Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
* Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Smith & Nephew (Allevyn® brand).

Study arm 2 (on top of standard of care):

* Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
* Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Mölnlycke Health care (Mepilex® brand).

Study arm 3 (standard of care):

* Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
* No silicone adhesive multilayer foam dressings will be applied on the skin sites of interest for this trial (sacrum, heel right/left, greater trochanter right/left).

Skin sites (restricted to sacrum, heel right/left, greater trochanter right/left) of patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will be assessed daily for a maximum period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. At risk for pressure ulcer development based on Braden risk assessment (Braden score ≤17).
2. Admitted to hospital within the previous 48 hours. Note: Not more than 25% of patients per site should be recruited at ICU wards.
3. Skin at sacrum is assessable and there is no clinically relevant incontinence- associated dermatitis (IAD*) or another skin condition that would be a contra-indication for the application of the devices under study, and there is no pressure ulcer category II or worse present.

   *clinically relevant IAD is defined as any of the 4 categories described in the publication http://users.ugent.be/~dibeeckm/globiadnl/nlv1.0.pdf
4. For at least 3 of the following 4 skin sites (heel left, heel right, greater trochanter left, greater trochanter right) one of the following two conditions should apply:

   - A study dressing can be applied as prevention of a pressure ulcer category II or worse at that skin site (there is no contra-indication)

   OR

   - There is already a pressure ulcer category II or worse at that skin site.
5. Written informed consent by the patient or his/her legal representative.

Exclusion Criteria:

1. Aged < 18 years.
2. The length of stay counting from first day of admission in one or (if the patient is transferred to another ward) more participating wards is < 7 days.
3. Both heels amputated
4. Previously known/documented allergy for substances used in the devices under study.
5. A clinical condition not allowing participation in a clinical study.
6. Participation in another interventional clinical trial.
7. Patients who exceptionally receive or are planned to receive a dressing for the prevention of pressure ulcers at sacrum, heels and trochanters based on best medical judgment and outside of the surgery setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1634 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, Principal Investigator — Ugent
Locations (8):
- Belgium (8):
  - OLV Aalst, Aalst
  - AZ Maria Middelares Ghent, Ghent
  - University of Ghent, Ghent
  - UZ Brussel, Jette
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - OLV van Lourdes Ziekenhuis Waregem, Waregem
  - AZ Sint-Elisabeth Zottegem, Zottegem

IPD SHARING:
Plan to Share IPD: Yes
Access will be granted to non-commercial researchers who provide a methodologically sound proposal for a relevant research questions. Relevance will be assessed by the Sponsor in collaboration with the Chief investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 12 months after publication for 5 years.
Access Criteria: To achieve aims in the approved proposal. Proposals should be directed to trials@KCE.fgov.be. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Beeckman D, Fourie A, Raepsaet C, Van Damme N, Manderlier B, De Meyer D, Beele H, Smet S, Demarre L, Vossaert R, de Graaf A, Verhaeghe L, Vandergheynst N, Hendrickx B, Hanssens V, Keymeulen H, Vanderwee K, Van De Woestijne J, Verhaeghe S, Van Hecke A, Savoye I, Harrison J, Vrijens F, Hulstaert F. Silicone adhesive multilayer foam dressings as adjuvant prophylactic therapy to prevent hospital-acquired pressure ulcers: a pragmatic noncommercial multicentre randomized open-label parallel-group medical device trial. Br J Dermatol. 2021 Jul;185(1):52-61. doi: 10.1111/bjd.19689. Epub 2020 Dec 28. PMID 33216969
- See also: Clinical Study Report — https://kce.fgov.be/sites/default/files/atoms/files/KCE-16012_Clinical%20Study%20Report_FINAL%2020201201.pdf
- See also: Study webpage — https://kce.fgov.be/en/kce16012-a-medical-device-trial-to-evaluate-the-use-of-a-silicone-adhesive-multilayer-foam-dressing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 68 wards in 8 hospitals (three university/teaching and five general hospitals) in Flanders, Belgium from February 2018 to December 2018.
  In total, 1680 participants were screened for eligibility and 1633 participants were randomised to one of the study arms. The number of participants randomised per study site varied between 64 and 287 (median 233).
  In the intention to treat (ITT) population 12.4% of patients were randomised in the ICU and 87.5% in non-ICUs.
Pre-assignment Details: 47 participants were excluded; 1 asked to have their data excluded from the analysis and 46 were not randomised.
Groups:
- Intervention Group 1 (on Top of Standard of Care): Allevyn® brand silicone adhesive multilayer foam dressings
  * Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Smith & Nephew (Allevyn® brand).
- Intervention Group 2 (on Top of Standard of Care): Mepilex® brand silicone adhesive multilayer foam dressings
  * Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Mölnlycke Health care (Mepilex® brand).
- Control Group (Standard of Care): * Patients at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * No silicone adhesive multilayer foam dressings will be applied on the skin sites of interest for this trial (sacrum, heel right/left, greater trochanter right/left).
Period: Overall Study
Arm/Group | Intervention Group 1 (on Top of Standard of Care) | Intervention Group 2 (on Top of Standard of Care) | Control Group (Standard of Care)
Started | 542 (All participants received at least 1 dressing) | 545 (One participant received one Allevyn® Life dressing (wrong brand by mistake), besides 13 Mepilex® Border on sacrum, (0.2%) All participants received at least 1 dressing) | 546 (No participants received dressings)
Completed (All participants completed the study however not all were included in the analysis.) | 534 | 532 | 539
Not Completed | 8 | 13 | 7
Not completed — Not included in analysis as assessed only once and no pressure ulcer or category 1 at any site | 8 | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group 1 (on Top of Standard of Care): Allevyn® brand silicone adhesive multilayer foam dressings
  * Participants at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Smith & Nephew (Allevyn® brand).
- Intervention Group 2 (on Top of Standard of Care): Mepilex® brand silicone adhesive multilayer foam dressings
  * Participants at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * Skin sites (restricted to sacrum, heel right/left and greater trochanter right/left) will be treated with silicone adhesive multilayer foam dressings by Mölnlycke Health care (Mepilex® brand).
- Control Group (Standard of Care): * Participants at risk for pressure ulcer category II, III, IV, Unstageable, and Deep Tissue Injury (DTI) development will receive standard pressure ulcer prevention strategies (as described in the hospital protocol) which include ongoing risk assessment, regular repositioning and skin care.
  * No silicone adhesive multilayer foam dressings will be applied on the skin sites of interest for this trial (sacrum, heel right/left, greater trochanter right/left).
- Total: Total of all reporting groups
Arm/Group | Intervention Group 1 (on Top of Standard of Care) | Intervention Group 2 (on Top of Standard of Care) | Control Group (Standard of Care) | Total
Number analyzed (Participants) | 542 | 545 | 546 | 1633
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.8 (12.3) | 79.4 (12.5) | 79.6 (11.7) | 79.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 320 | 302 | 319 | 941
  Male | 222 | 243 | 227 | 692
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Ward type at study start [Count of Participants; unit: Participants]
  ICU | 65 | 67 | 71 | 203
  Non-ICU | 477 | 478 | 475 | 1430
Total Braden score (at Baseline) [Mean (Standard Deviation); unit: units on a scale] — The Braden Scale for Predicting Pressure Sore Risk (Bergstrom, Braden, Laguzza & Holman, 1987) is composed of six sub-scales that reflect sensory perception, skin moisture, activity, mobility, friction and shear, and nutritional status. Each sub-scale is scored from 1-3 or 4, for total scores that range from 6-23. A lower Braden Scale Score indicates a lower level of functioning and, therefore, a higher level of risk for pressure ulcer development. In this study a cut-off of <= 17 was used for being at risk of pressure ulcer development.
  units on a scale | 13.0 (2.3) | 13.1 (2.5) | 13.0 (2.3) | 13.0 (2.4)
BMI (kg/m²) [Count of Participants; unit: Participants]
  Underweight (<18.5) | 44 | 53 | 39 | 136
  Normal weight (18.5-25.0) | 234 | 249 | 258 | 741
  Overweight (25.0-30.0) | 161 | 163 | 162 | 486
  Obese (>30.0) | 103 | 80 | 87 | 270
Diabetes [Count of Participants; unit: Participants]
  No diabetes | 419 | 427 | 412 | 1258
  Diabetes | 123 | 118 | 134 | 375
Surgery since admission [Count of Participants; unit: Participants] — Participants who had had surgery since admission to hospital (and prior to consent/randomization in the study).
  Participants
    No surgery | 484 | 486 | 489 | 1459
    Surgery | 58 | 59 | 57 | 174

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed a New Pressure Ulcer Category 2 or Worse on Sacrum, Heels or Greater Trochanter
Description: The number of participants who developed at least one new pressure ulcer of category 2 or worse on sacrum, heels or greater trochanter as judged onsite, during the study period (maximum 14 days).
  Patients in experimental groups 1 and 2 were pooled as the treatment group and compared to the control group (in the intention to treat population (n=1605)
  Note: The International NPUAP/EPUAP Pressure Ulcer Classification System (National Pressure Ulcer Advisory Panel (2014)) distinguishes four categories of pressure ulcers: non-blanchable erythema of the intact skin (category I), partial thickness loss of dermis (category II), full thickness tissue loss (category III) and full thickness tissue loss with exposed bone, tendon or muscle (category IV). Also unstageable pressure ulcers and deep tissue injuries can be recognised. https://npiap.com/
Time Frame: assessment during 14 days
Population: Intention to treat population (n=1605)
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Group (Defined in Protocol as Pooled Intervention Group 1 and Intervention Group 2): Participants in intervention groups 1 and 2
  * were cared for on the available support surfaces of the hospital (mattresses, cushions) for the duration of their hospital stay.
  * received standard pressure ulcer prevention strategies (as described in the hospital protocol) which included ongoing risk assessment, regular repositioning and skin care.
  * Silicone adhesive multilayer foam dressings were applied on dry intact skin on sacrum, heel right/left, greater trochanter right/left, in addition to standard pressure ulcer prevention.
  * The maximum treatment duration was 14 days
- Control Group: Participants in control group
  * were cared for on the available support surfaces of the hospital (mattresses, cushions) for the duration of their hospital stay.
  * received standard pressure ulcer prevention strategies (as described in the hospital protocol) which included ongoing risk assessment, regular repositioning and skin care.
  * No silicone adhesive multilayer foam dressings were applied
  * The maximum study duration was 14 days
Arm/Group | Treatment Group (Defined in Protocol as Pooled Intervention Group 1 and Intervention Group 2) | Control Group
Number analyzed (Participants) | 1066 | 539
Participants | 43 | 34
Statistical Analysis 1: Comparison: Treatment Group (Defined in Protocol as Pooled Intervention Group 1 and Intervention Group 2) vs Control Group; Test type: Superiority; p = 0.04, Cochran-Mantel-Haenszel — controlled for type of ward (ICU/Non-ICU); Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.41 to 0.99]

2. Other Pre Specified Outcome: Number of Participants Who Developed a New Pressure Ulcer Category 2 or Worse on Sacrum
Description: The number of participants who developed at least one new pressure ulcer of category 2 or worse on sacrum as judged onsite, during the study period (maximum 14 days).
Time Frame: maximum treatment or study period 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group (Defined in Protocol as Pooled Intervention Group 1 and Intervention Group 2) | Control Group
Number analyzed (Participants) | 1066 | 539
Participants | 30 | 26

3. Other Pre Specified Outcome: Number of Participants Who Developed a New Pressure Ulcer Category 2 or Worse on Any Heel
Description: The number of participants who developed at least one new pressure ulcer of category 2 or worse on any heel as judged onsite, during the study period (maximum 14 days).
Time Frame: maximum treatment or study period 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group (Defined in Protocol as Pooled Intervention Group 1 and Intervention Group 2) | Control Group
Number analyzed (Participants) | 1066 | 539
Participants | 15 | 10

4. Other Pre Specified Outcome: The Number of Participants Who Developed a New Pressure Ulcer Category 2 or Worse on Any Trochanter
Description: The number of patients who developed at least one new pressure ulcer of category 2 or worse on any greater trochanter as judged onsite, during the study period (maximum 14 days).
Time Frame: maximum treatment or study period 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group (Defined in Protocol as Pooled Intervention Group 1 and Intervention Group 2) | Control Group
Number analyzed (Participants) | 1066 | 539
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: They will be recorded between the first usage of the study dressings and the last study related intervention for that patient for Adverse Device Events (ADEs) (usually maximum 14 days) and till 30 days after last study related intervention for SADEs/MDIs.
Description: Only ADEs, SADEs (i.e. AE/SAEs considered related to intervention, the study dressings and their application) and device deficiencies were recorded. The safety population (n=1077) was calculated after exclusion of participants in the ITT population who wanted their data excluded (n=1), who were not randomized (n=46), did not receive at least one dressing (n=10) or received only standard of care (n=546).
  Skin under the dressings was inspected every day.
Arm/Group | Intervention Group 1 (on Top of Standard of Care) | Intervention Group 2 (on Top of Standard of Care)
All-Cause Mortality (participants affected / at risk) | 27/539 | 23/538
Serious Adverse Events (participants affected / at risk) | 0/539 | 0/538
Other Adverse Events (participants affected / at risk) | 16/539 | 12/538
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group 1 (on Top of Standard of Care) (N=539) | Intervention Group 2 (on Top of Standard of Care) (N=538)
Pressure ulcer development (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) — Note: two of these pressure ulcers were category 1 and one was category 2
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Blister formation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Exacerbates athlete's foot (Infections and infestations) | 0 (0) | 1 (1)
Mechanical skin injuries (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
Patient fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pain at sacrum (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Performance and detection bias may have occurred because patients, caregivers and study personnel could not be blinded to the study procedures/devices. All study nurses were trained, and for most hospitals wound care teams were involved when a PU occurred, further strengthening the correct identification of skin injuries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03442777/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT03442777/SAP_001.pdf